CLINICAL TRIAL: NCT02367560
Title: Calcific Tendinitis: Comparing Minimally Invasive Modalities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lakehead University (Other)
Responsible Party: Principal Investigator, Jubin Payandeh, Orthopedic Surgeon, Assistant Professor, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP-336-10202014
Record Dates: First submitted 2015-01-21; First posted 2015-02-20 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Calcific Tendinitis
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Methylprednisolone Acetate; Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NDSSI (Active Comparator): Participants in this arm of the trial will be referred for Needle decompression with subacromial steroid (Depo medrol) injection (NDSSI) as their treatment for calcific tendinitis
  Interventions: Procedure: Needle decompression; Drug: Depo medrol
- SWT (Active Comparator): Participants in this arm of the trial will be referred for Shockwave therapy (SWT) using an Ultrasound device, delivered by a physiotherapist, as their treatment for calcific tendinitis
  Interventions: Procedure: Shockwave therapy; Device: Ultrasound device

INTERVENTIONS:
Procedure: Needle decompression — Direct manipulation of calcium deposits in the shoulder with a needle to fragment the deposit performed by a radiologist.
  Arms: NDSSI
Procedure: Shockwave therapy — A physiotherapist performs the shockwave therapy procedure. Treatment is completed in 4 weekly sessions. Treatment involves applying soundwaves directly to the affected shoulder area using an ultrasound device.
  Arms: SWT
Drug: Depo medrol — Subacromial steroid injection (40 mg depo medrol) is given to the patient to limit irritation following needle decompression.
  Other Names: methylprednisolone acetate Injectable Suspension
  Arms: NDSSI
Device: Ultrasound device — Ultrasound device is applied directly to the shoulder at 0.2 mJ/mm2.
  Arms: SWT

SUMMARY:
Calcific tendinitis is a common and challenging problem in the orthopedic surgeon's office. The chronic and variable course of the condition can lead to dissatisfaction with conservative management. Current standard of care at the Thunder Bay Regional Health Sciences Centre is referral for treatment by either needle decompression therapy by a radiologist or shockwave therapy by a physiotherapist. The purpose of this study is to compare the efficacies of these treatment options.

DETAILED DESCRIPTION:
Calcific tendinitis is a common and challenging problem in the orthopedic surgeon's office. The chronic and variable course of the condition can lead to dissatisfaction with conservative management. Current guidelines recommend conservative management initially and failing this, a variety of minimally invasive options exist. These include subacromial steroid injection (SSI), needle decompression (ND), and Shock wave therapy (SWT).

Few trials of these methods exist, but generally a benefit is seen with all minimally invasive methods. Most promising results have occurred with needle decompression and shockwave therapy. To date, no direct trials comparing SWT and ND have been published.

The purpose of this trial is to preliminarily establish the comparative efficacies of NDSSI and SWT using a number of outcome measures. Secondarily, the investigators aim to determine prognostic factors for success of minimally invasive therapies. The results of this study will serve as a foundation for more rigorous trials in this area.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of symptomatic calcific tendinitis of the shoulder
* Seeking treatment for diagnosis
* ≥ 18 years of age

Exclusion Criteria:

* Pre-existing diagnosis of rotator cuff tear or arthropathy
* Previous minimally invasive or surgical therapy
* Systemic Inflammatory disease
* Blood dyscrasia
* Peripheral neuropathy
* Active Workplace Safety & Insurance Board (WSIB) claim for shoulder injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change of Range of Motion | Baseline, 3 months, 1 year
  The change in a Participant's Range of Motion as measured by a goniometer (Passive Range of Motion [PROM] and Assistive Range of Motion [AROM]) from baseline to 3 months and 1 year.
Change of Western Ontario Rotator Cuff (WORC) score | Baseline, 3 months, 1 year
  Change in a participant's WORC scores from baseline to 3 months and 1 year. WORC is a condition-specific outcome tool for people with rotator cuff disorder. A total score for each domain is calculated (Physical Symptoms/600; Sports and Recreation/400; Work/400 and Lifestyle/400;Emotions/400) and the total score for the domains is summed for an aggregate score out of 2100.
Change of Gartland Classification of X-ray | Baseline, 3 months, 1 year
  The change in radiographic resolution as measured by the Gartland Classification scale (1-4) from baseline to 3 months and 1 year.

SECONDARY OUTCOMES:
The change in overall health as measured by the SF-8 | Baseline, 3 months, 1 year
  The change in SF-8 from baseline to 3 months and 1 year will be measured. SF-8 is a comprehensive health survey which calculates a score for health in 8 dimensions and as a summed result.

CONTACTS AND LOCATIONS:
Overall Officials: Jubin Payandeh, MD, Principal Investigator — Thunder Bay Regional Health Sciences Centre
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No